CLINICAL TRIAL: NCT03391726
Title: CART-19 Cells For Patients With Relapsed or Refractory B-cell Lymphoma
Brief Title: CART-19 Cells for R/R B-cell Lymphoma
Acronym: CCFRRBL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Jianda Hu, Director of the department of Hematology, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-19-01
Record Dates: First submitted 2017-12-30; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Relapsed or Refractory B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): CART-19 cells treat
  Interventions: Other: CART-19 cells

INTERVENTIONS:
Other: CART-19 cells — CART-19 cells treat

SUMMARY:
Relapsed/Refractory B Cell Lymphoma is a challenge to be treated, however,CART-19 cells could be very promosing. This study aims to assess the safety and toxicity of CART-19 cells for patients with relapse or refractory B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged between 1-65 years
* Patients with relapse/refractory B-cell lymphoma
* Cardiac: Left ventricular ejection fraction ≥ 50%
* Adequate renal and hepatic function
* Performance status: Karnofsky ≥ 70%

Exclusion Criteria:

* Pregnant or lactating females.
* Any co-morbidity precluding the administration of CART-19 cells.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 1 year

SECONDARY OUTCOMES:
Adverse events that are related to treatment | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China